CLINICAL TRIAL: NCT05806372
Title: Biomarkers of Maternal Cardio-vascular Dysfunction in Pregnancies Complicated by Hypertensive Disorders of Pregnancy
Brief Title: Biomarkers of CVD Dysfunction in Hypertensive Disorders of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 29/22
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Diseases; Pregnancy
Keywords: Cardiomyocytes; microRNA,; hypertensive disorders of pregnancy
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — sera of women that experienced HDP with and without FGR will be used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HDP with FGR: Evaluation of sera and ultrasound data on fetal growth and Doppler velocimetry in women with HDP and fetal growth restriction.
- HDP without FGR: Evaluation of sera and ultrasound data on fetal growth and Doppler velocimetry in women with HDP and without fetal growth restriction.
- Normotensive: Evaluation of sera and ultrasound data on fetal growth and Doppler velocimetry in normotensive women.

SUMMARY:
Profound and concomitant cardiovascular hemodynamic changes, necessary to support fetoplacental development and its increasing supply demands, occur during a physiological pregnancy characterized by an increase in cardiac output, heart rate and plasma volume, and fall in vascular resistance and blood pressure. The result of these changes is a volume overload that will lead to a compensatory transient left ventricular eccentric hypertrophy. This, together with the pro-inflammatory state typical of pregnancy, represents the pregnancy as a stress-test for the maternal cardiovascular system. Pregnancies complicated by hypertensive disorders of pregnancy (HDP), particularly those with early onset and/or complicated by intrauterine fetal growth restriction (FGR), are characterized by a cardiovascular maladaptation. Women who experienced HDP in pregnancy, especially pre-eclampsia (PE), more often develop later in life ischemic heart disease, hypertension and stroke, obesity, dyslipidemia, and end-stage renal disease.

Regardless its clinical impact, very little knowledge is available on the mechanisms by which PE could lead to cardiovascular disease (CVD), and, especially, to heart failure after pregnancy. Preliminary results suggest a cross-talk between pregnancy-induced biomarkers and cardio-vascular system. Particularly, cultures of neonatal rat cardiomyocytes and fibroblasts were used to investigate the role of the serum of women with HDP in regulating their proliferation. 5-ethynyl-2'-deoxyuridine (EdU) was administered to label DNA synthesis in proliferating cells. After 3 days of in vitro culture, EdU incorporation was analyzed upon immunofluorescence staining using specific antibodies by high content microscopy. A possible protective effect exerted by the selected sera against apoptosis was evaluated, as well, by Caspase activation. Moreover, the effect of cardiomyocytes and fibroblasts proliferation and apoptosis on maternal hemodynamic parameters was evaluated using median regression models. These data show that the serum of women with HDP triggers a net increase in the percentage of proliferating cardiomyocytes compared to controls. Moreover, there were relationship between cardiomyocytes and fibroblasts proliferation and maternal hemodynamics parameters thus, supporting the hypothesis that the serum of women with HDP may contain factors capable of stimulating cardiac cells in response to the cardiovascular stress-test

ELIGIBILITY:
Inclusion Criteria:

CASES:

1. Pregnant women affected by HDP
2. Women ≥18 years old
3. Women able to give an informed consent

CONTROLS

1. Uneventful pregnancy of women ≥18 years old
2. Women able to give an informed consent

Exclusion Criteria:

1. No informed consent
2. Women <18 years old
3. Presence of other maternal pathologies as viral disease, diabetes
4. Fetal chromosomal/structural anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Singleton pregnant women between 24 and 40 gestational weeks with HDP (with and without fetal growth disorder) and normotensive (controls)
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of biomarkers predicting cardiomyocyte hypertrophy and fibroblast proliferation | During pregnancy, at the time of HDP diagnosis
  By exploiting the availability of a library of viral vectors encoding for the whole secretome (about 1200 secreted proteins) and the whole miRNAome (about 2000 human microRNAs) a high throughput screening will be carried out to identify molecules able to control the viability, proliferation and cell size of both primary cardiomyocytes and cardiac fibroblasts. Data mining methods for multi-target prediction, such as ensembles of predictive clustering trees, will be used to correlate multiple independent variables (e.g., potential biomarkers) to the multiple clinical outcomes (indices of cardio-vascular dysfunction measured by echocardiography).
Number of biomarkers predicting cardiomyocyte hypertrophy and fibroblast proliferation | 24 months post-partum
  By exploiting the availability of a library of viral vectors encoding for the whole secretome (about 1200 secreted proteins) and the whole miRNAome (about 2000 human microRNAs) a high throughput screening will be carried out to identify molecules able to control the viability, proliferation and cell size of both primary cardiomyocytes and cardiac fibroblasts. Data mining methods for multi-target prediction, such as ensembles of predictive clustering trees, will be used to correlate multiple independent variables (e.g., potential biomarkers) to the multiple clinical outcomes (indices of cardio-vascular dysfunction measured by echocardiography).

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Stampalija, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided